CLINICAL TRIAL: NCT06970444
Title: The Effect of Transcutaneous Auricular Vagal Nerve Stimulation on Auditory Processing Abilities in Healthy Individuals
Brief Title: taVNS Effect on Central Auditory Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ayberk Aydın Tunc, Audiologist, M.Sc., Medipol University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MedipolU-Aud-01
Record Dates: First submitted 2025-03-20; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Central Auditory Disease; Auditory Processing Disorder, Central; Auditory Processing Disorders; Vagus Nerve Stimulation
Keywords: central auditory processing; transcutaneous auricular vagus nerve stimulation; central auditory processing disorder; aural rehabilitation
MeSH Terms: conditions — Auditory Diseases, Central; Language Development Disorders; Auditory Perceptual Disorders

STUDY DESIGN:
Intervention Model Description: We evaluate the Central Processing skills before and after the stimulations (real and sham stimulation). This was a non-invasive stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- taVNS Group (Experimental): The group which recieved taVNS stimulation through their left ear
  Interventions: Device: transcutaneous auricular vagus nerve stimulation (taVNS)
- Sham (Placebo) g,Group (Sham Comparator): control group received sham stimulation with the stimulator closed and electrodes placed in their left ear
  Interventions: Other: Sham device

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation (taVNS) — Transcutaneous auricular vagus nerve stimulation (taVNS) is an emerging non-invasive therapy that modulates brain activity by delivering electrical impulses to the auricular branch of the vagus nerve at the outer ear (Badran et al., 2018). taVNS subsequently stimulates the nucleus of tractus solitarius via the afferent vagus nerve fibers. The nucleus solitarius sends outputs to the hypothalamus, which is critical for sensory processing, including auditory processing, and also activates various brain regions, including the locus coeruleus, resulting in the release of neurotransmitters such as norepinephrine and serotonin, which are involved in neural plasticity and cognitive function, which is important for CAP. Another theory for taVNS effects is the release of gamma-aminobutyric acid (GABA), an inhibitory neurotransmitter, which may further help to balance abnormal neural activity in auditory circuits.
  Arms: taVNS Group
Other: Sham device — the control group received sham stimulation with the stimulator closed and electrodes placed in their left ear
  Arms: Sham (Placebo) g,Group

SUMMARY:
The behavioral effects of vagus nerve stimulation (VNS) and observed activation in the auditory cortex with transcutaneous auricular VNS (taVNS) raise questions about their potential impact on auditory processing. This study aims to investigate whether taVNS, which has not been studied in the context of central auditory processing (CAP), has any effects on CAP.

DETAILED DESCRIPTION:
Experimental procedure First, the participants were made to sign the 'Informed Volunteer Consent Form'. Then, the MoCA test was applied, and pure tone audiometry test was performed on those who scored 21 or above and were determined to have normal cognitive abilities. After air and bone conduction pure tone thresholds were determined, speech reception thresholds with three-syllable phonetically balanced words and Speech Discrimination Scores (SDS) with monosyllabic phonetically balanced words were measured. Participants with normal hearing were included in the study. Central Auditory Processing (CAP) tests, Frequency Patterns Test (FPT) and Duration Patterns Test (DPT) were applied to the participants in the study group separately for each ear, and the current situation in the CAP evaluation was recorded. Then, taVNS was applied to left ear for 15 minutes with a biphasic, square stimulus with a pulse width of 250 µs, a stimulus at the sensor threshold level and a frequency of 20 Hz. The control group received sham stimulation with the stimulator closed and electrodes placed. After the stimulations, CAP tests were repeated for each ear separately. Differences between the study and control groups were examined. The application was performed in a dimly lit, sound-insulated double-walled cabin (a sound-insulated room in accordance with Industrial Acoustics 18 Company [IAC] standards), while sitting in a comfortable chair. The audio file was opened from the desktop computer and sent via the aux cable to the clinical audiometer device (AC40 Clinical Audiometer). The participant listened to the sound through supraaural headphones (TDH39).

70 healthy participants with 140 ears were included in the study. Participants were 18-40 years old. 40 people; 20 females (23,20±2,35 mean of years) were included in the study group with active taVNS and 30 people; 15 females (23,30±3,48 mean of years) were included in the control group. All participants were native Turkish speakers with normal cognitive conditions and hearing which has been demonstrated by routine tests. Further inclusion criteria were: age 18-40 years, normal CAP performance. The age range of the study was determined by taking into account that CAP skills decrease with increasing age. In order to eliminate heterogeneity, male-female balance was taken into account. As the effect of hemispheric lateralization, those with left hand dominance had differences in language skills and spatial attention, and in verbal and non-verbal behavioral tasks, compared to those with right hand dominance, only individuals with right hand dominance were included in the study, taking into account that it may affect the test results. Musical training is an important factor in FPT performance as it provides better frequency discrimination perception. Therefore, individuals with a professional music background were not included in the study, as it was thought that it could affect brain organization and cause differences in test results.

To evaluate cognitive functions, the MoCA test, was applied to the participants. Who scored 21 or above were determined to have normal cognitive abilities.

To confirm that the hearing abilities of the individuals participating in the study were normal, a pure tone and speech audiometry test and FPT-DPT test batteries were performed using the Interacoustic AC40 (Denmark) audiometer device. The hearing thresholds of octave band frequencies thresholds of 250 Hz to 8000 Hz were 25 dB or lower were considered normal.

FPT and DPT were applied to the participants, respectively. During or at the end of the tests, breaks were taken according to the participants' wishes so that they could focus.

FPT is a test battery developed to evaluate temporal sequencing ability, which is one of the subcategories of temporal processing. In our study, for FPT, an audio -mp3- file based on the parameters determined by Musiek was applied. The high frequency sound used as test stimulus frequencies was determined as 1122 Hz, and the low frequency sound was determined as 880 Hz. The length of the stimulus period was determined as 200 ms, and the inter-stimulus interval was 150 ms. There is a 10 ms rise-fall time between the stimuli. There were six possible combinations of tones (Low-Low-High (LLH), LHL, LHH, HLH, HLL and HHL). Participants were asked to verbally rank the sounds they heard according to their frequency and order of occurrence, and several stimulus sets were presented for trial purposes before the test, not to be included in the scoring. The test started when the participant indicated that she/he was ready. Stimuli were presented at 60 dB HL through TDH-39 over-ear headphones. Participants were presented with a total of 50 sets of stimuli, 25 triple stimuli for each ear, and FPT scores were calculated as a percentage for both ears separately.

It is a test set that measures another temporal sequencing skill known as DPT. In our study, sound recording for DPT was made using an audiometer in line with the criteria determined by Musiek. Stimuli were presented at a frequency of 1000 Hz. Long duration sounds were determined as 500 ms, and short duration sounds were determined as 250 ms. There was a 10 ms rise and fall time between stimuli. The interstimulus interval was set at 300 ms. There were six possible combinations of tones (Long-Long-Short (LLS), LSS, LSL, SLL, SSL, SLS). Participants were asked to verbally rank the sounds they heard according to their duration and the order in which they were presented, and stimulus sets were presented for trial purposes not to be included in the scoring. Before the test began, participants were asked to indicate their readiness. Stimuli were presented in a total of 50 sets, 25 triple stimuli for each ear, at 60 dB HL level, and separate DPT scores were calculated for both ears.

FPT and DPT allow participants to express some of the stimulus patterns presented to them in reverse. In the literature, 2 score types have been defined in which this situation is accepted as a right or wrong. In our study, scoring was done according to both score types.

These score types are listed below:

Rev Plus: Score type calculated by accepting the reversed patterns as correct that we mentioned as "Rev." in the tables.

Rev Minus: Score type calculated by accepting the reversed patterns as incorrect.

taVNS parameters After the first CAP evaluations of the participants in the study group, taVNS was applied via VAGUSTIM TENS (Vagustim Health Technologies, San Francisco, CA, USA) device. Stimulating electrodes were placed on the inner surface of the left ear between the tragus and concha (Figure2). Ultrasound gel was applied to the electrodes during placement to increase electrical conduction. Then, stimulation parameters adjusted and stimulation started. The stimulation amplitude increased gradually, with the guidance of the participants, at a comfortable level (sensory treshold level), where the stimulation was felt but did not cause pain or discomfort. Stimulation time was set as 15 minutes. Stimulation duration was limited to 15 minutes to prevent possible side effects like hypotension, dizziness, etc.

Stimulus parameters used when applying taVNS to the left ear: In the study of Peng et al., the stimulus parameters proven by f-MRI to create activity in the auditory cortex were taken as a reference. A biphasic modified square stimulus with a pulse width of 250 µs. Electric current amplitude threshold was adjusted according to participant tolerance. The stimulation frequency was kept at 20 Hz, which is known to activate nerve fibers.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-40 years old
* Having a score of 21 or above on the MoCA test
* Having a normal range on the bilateral pure tone audiometry test
* Having no problems on any scanner
* Having no professional music background
* Having right hand dominance
* Having no contraindication to T-a-VNS

Exclusion Criteria:

* Peripheral hearing disorders
* Professional music history
* Physical and emotional disorders that may affect the test results
* Left-hand dominance
* Persons in whom the use of T-a-VSU is contraindicated

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Frequency Patterns Test (FPT) | Immediately before and after the stimulation (totally: 30 min)
  FPT is a test battery developed to evaluate temporal sequencing ability, which is one of the subcategories of temporal processing. In our study, for FPT, an audio -mp3- file based on the parameters determined by Musiek was applied. The high frequency sound used as test stimulus frequencies was determined as 1122 Hz, and the low frequency sound was determined as 880 Hz. The length of the stimulus period was determined as 200 ms, and the inter-stimulus interval was 150 ms. There is a 10 ms rise-fall time between the stimuli. There were six possible combinations of tones (Low-Low-High (LLH), LHL, LHH, HLH, HLL and HHL). Participants were asked to verbally rank the sounds they heard according to their frequency and order of occurrence, and several stimulus sets were presented for trial purposes before the test, not to be included in the scoring.
Duration Patterns Test (DPT) | Immediately before and after the stimulation (totally: 30 min)
  It is a test set that measures another temporal sequencing skill known as DPT (Musiek et al., 1990). In our study, sound recording for DPT was made using an audiometer in line with the criteria determined by Musiek. Stimuli were presented at a frequency of 1000 Hz. Long duration sounds were determined as 500 ms, and short duration sounds were determined as 250 ms. There was a 10 ms rise and fall time between stimuli. The interstimulus interval was set at 300 ms. There were six possible combinations of tones (Long-Long-Short (LLS), LSS, LSL, SLL, SSL, SLS). Participants were asked to verbally rank the sounds they heard according to their duration and the order in which they were presented, and stimulus sets were presented for trial purposes not to be included in the scoring. Before the test began, participants were asked to indicate their readiness. Stimuli were presented in a total of 50 sets, 25 triple stimuli for each ear, at 60 dB HL level, and separate DPT scores were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ayberk Aydin Tunç, Master of Science, Principal Investigator — Istanbul Medipol University, Audiology Department
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Taeye L, Vonck K, van Bochove M, Boon P, Van Roost D, Mollet L, Meurs A, De Herdt V, Carrette E, Dauwe I, Gadeyne S, van Mierlo P, Verguts T, Raedt R. The P3 event-related potential is a biomarker for the efficacy of vagus nerve stimulation in patients with epilepsy. Neurotherapeutics. 2014 Jul;11(3):612-22. doi: 10.1007/s13311-014-0272-3. PMID 24711167
- [Background] Peng L, Mu K, Liu A, Zhou L, Gao Y, Shenoy IT, Mei Z, Chen Q. Transauricular vagus nerve stimulation at auricular acupoints Kindey (CO10), Yidan (CO11), Liver (CO12) and Shenmen (TF4) can induce auditory and limbic cortices activation measured by fMRI. Hear Res. 2018 Mar;359:1-12. doi: 10.1016/j.heares.2017.12.003. Epub 2017 Dec 24. PMID 29305037
- [Background] Musiek, F. E. (2002). The frequency pattern test: A guide. Hearing Journal, 55(6), 58. https://doi.org/10.1097/01.HJ.0000293280.99394.DD
- [Background] Musiek FE. Frequency (pitch) and duration pattern tests. J Am Acad Audiol. 1994 Jul;5(4):265-8. PMID 7949300